CLINICAL TRIAL: NCT07323472
Title: Analysis of Respiratory Drive Activation, Ventilation, and Pulmonary Aeration Resulting From Body Lateralization in Critically Ill Patients Under Mechanical Ventilation
Brief Title: Body Lateralization and Its Effects on Respiratory Drive, Ventilation, and Pulmonary Aeration in Critically Ill Patients
Acronym: LATLUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Shirley Lima Campos, Principal Researcher, University of Pernambuco
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LATLUNG; 92079725.0.0000.5208 (Other: Research Ethics Committee on Human Research, Federal University of Pernambuco - Recife Campus (UFPE/Recife))
Record Dates: First submitted 2025-11-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care Units (ICUs)
Keywords: Automatic lateralization therapy; Critical illness; Continuous lateral rotation; Electrical impedance tomography; Surface electromyography; Respiratory muscles
MeSH Terms: conditions — Critical Illness | interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study with a non-randomized physiological interventional design in a single group of critically ill adult patients under mechanical ventilation. Each participant will undergo all intervention conditions, including different body lateralization angles (0°, 15°, 30°) with Automatic Lateralization Therapy with and without Flow Bias. Repeated measures will include respiratory drive, ventilation, and pulmonary aeration assessed by P0.1, estimated Pmus, sEMG, EIT, and ultrasound, allowing each participant to serve as their own control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Apart from the participants and the researchers responsible for data analysis, no other role is blinded in the study.
  The researchers responsible for carrying out the interventions and conducting the study are not blinded to the intervention conditions.
  Blinding is applied only to:
  * Participants: sedated and, therefore, unaware of the intervention received.
  * Researchers responsible for data analysis: blinded to the intervention conditions during the evaluation of physiological and ventilatory parameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supine Positioning (Active Comparator): Participants will remain in supine position with 30° head elevation. No lateralization therapy is applied.
  Interventions: Other: Supine Positioning
- Automatic lateralization therapy (Active Comparator): Participants will undergo continuous lateral positioning on an automated bed, with automatic angle and time adjustments. The second sequence will be combined with the Flow Bias intervention.
  Interventions: Other: Automatic Lateralization Therapy

INTERVENTIONS:
Other: Automatic Lateralization Therapy — During this phase of analysis and intervention related to lateral positioning, patients will be maintained on a Multicare bed (LINET) and subjected to personalized lateral positioning based on the morphofunctional pattern detected by electrical impedance tomography. This positioning will be performed using automatic lateralization therapy, programmed for unilateral or bilateral application, continuously alternating between angles of 0°, 15°, and 30°, maintained for 20 minutes at each position. The procedure will be conducted in two sequences, with the second sequence combined with the Flow Bias intervention. At each angle, data will be collected on hemodynamic monitoring, respiratory drive, respiratory mechanics, regional distribution of ventilation and aeration, and gas exchange.
  Other Names: Continuous lateral positioning; Automatic patient positioning; Continuous lateral rotation therapy; Lateral rotation therapy; Continuous rotational therapy; Kinetic bed therapy; Lateral change Positioning; Automated lateral rotation; Rotating bed; Automatic lateral therapy; Kinetic Therapy; Automated Lateral Rotation Therapy
  Arms: Automatic lateralization therapy
Other: Supine Positioning — During this analysis phase, patients will be positioned on a Multicare bed (LINET) in the dorsal decubitus position with the head of the bed elevated to 30°. Data will be collected on hemodynamic monitoring, respiratory drive, respiratory mechanics, degree of lung involvement, regional distribution of ventilation and aeration, and gas exchange.
  Other Names: Supine; Semi-recumbent position; Recumbent position; Dorsal decubitus; Conventional supine care
  Arms: Supine Positioning

SUMMARY:
The goal of this quasi-experimental study is to investigate how different body positions, performed through Automatic Lateralization Therapy, affect respiratory drive, ventilation, and pulmonary aeration in critically ill adult patients under mechanical ventilation. The main questions this study aims to answer are:

* Does Automatic Lateralization Therapy, modify respiratory drive, as measured by P0.1, estimated Pmus, and sEMG of the diaphragm and parasternal muscles?
* Is there an association between respiratory drive, ventilation, and pulmonary aeration measured by Electrical Impedance Tomography (EIT) in different body positions promoted by Automatic Lateralization Therapy ?

Does combining Automatic Lateralization Therapy, with Flow Bias improve physiological and functional outcomes compared to Automatic Lateralization Therapy, without Flow Bias?

Participants will:

* Be positioned in different lateralization strategies using Automatic Lateralization Therapy, while under mechanical ventilation;
* Have respiratory parameters and ventilation images assessed by EIT and sEMG;

Participate only during their ICU stay, with no need for additional visits after discharge.

DETAILED DESCRIPTION:
Detailed Description:

Critically ill patients under mechanical ventilation frequently develop respiratory complications due to immobility and altered pulmonary mechanics. Automatic Lateralization Therapy has emerged as a promising physiologic intervention to optimize ventilation and reduce respiratory dysfunction in this population. However, its effects on respiratory drive activation remain poorly understood.

Objective:

To evaluate the effects of body lateralization on respiratory drive activation, ventilation, and pulmonary aeration in mechanically ventilated critically ill patients.

Methods and Design:

This is a quasi-experimental, non-randomized physiological intervention study conducted in a controlled ICU environment, following the TREND 2025 Statement Checklist for transparent reporting of non-randomized evaluations. Automatic Lateralization Therapy will be applied with and without Flow Bias, using progressive body tilt angles (0°, 15°, and 30°). Positioning strategies will be personalized based on Electrical Impedance Tomography (EIT) findings to ensure optimal lung recruitment and safety.

Collected data will include:

Clinical and physiological parameters such as respiratory drive (P0.1, estimated Pmus),

Diaphragm and parasternal muscle activity via surface electromyography (sEMG),

Ventilatory mechanics and gas exchange,

Pulmonary aeration and regional ventilation distribution assessed by EIT,

Additional monitoring by lung ultrasound to confirm aeration patterns.

The investigator performing the physiological data analysis will be blinded to the intervention group to minimize bias. Cardiorespiratory safety (e.g., hemodynamic stability, oxygenation) and adverse events will be monitored throughout all procedures.

Expected Outcomes:

The study aims to provide insights into whether body lateralization through Automatic Lateralization Therapy, modulates respiratory drive and improves ventilation efficiency in critically ill patients. It is hypothesized that combining Automatic Lateralization Therapy, with Flow Bias will enhance pulmonary expansion, respiratory drive activation, and gas exchange efficiency compared to Automatic Lateralization Therapy, alone, while maintaining patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes will be included;
* Aged ≥ 18 years;
* BMI 18-35 kg/m²;
* Under invasive mechanical ventilation via orotracheal tube for ≥ 24 hours and expected to remain on mechanical ventilatory support for at least 48 hours;
* Sedated (Richmond Agitation-Sedation Scale [RASS] -1 to -4);
* Well adapted to protective ventilation strategies in VCV or PSV modes;
* Presenting neural respiratory drive evidenced by a drop in Delta Pocc and/or the presence of assisted cycles;
* Hemodynamically stable (mean arterial pressure between 60-120 mmHg, systolic arterial pressure between 90-180 mmHg, diastolic arterial pressure between 60-100 mmHg, and heart rate between 50-150 bpm) with or without vasoactive drugs at the time of data collection (> 0.1 to 0.3 mcg/kg/min);
* Respiratory stability, no use of accessory muscles and target SpO₂ achieved;
* No indication for nebulization or heated humidification at the time of collection;
* Positive tolerance test for lateral decubitus positioning;
* Chest circumference of 78-87.9 cm (XS), 88-99.9 cm (S), or 100-111.9 cm (M).

Exclusion Criteria:

* Patients presenting medical restrictions to body repositioning, or to the use of EIT or sEMG;
* Those in therapeutic failure;
* Individuals with spinal cord injury, brain injury, or stroke with a history of functional loss and respiratory impairment prior to hospitalization;
* Neurological diseases affecting respiratory myoelectric conduction;
* History of postural deformities, diaphragmatic abnormalities, or colostomy bag;
* Unstable fracture (lower or upper limbs in proximal regions or thorax);
* Pleural effusion requiring drainage;
* Presence of drains in the thoracic and/or abdominal regions;
* Unstable intracranial pressure;
* Pregnant patients;
* Immediate postoperative period of orthopedic surgeries;
* Use of mucolytics;
* Open ventriculostomy for drainage;
* Uncontrolled agitation;
* Pacemaker or implantable cardioverter-defibrillator;
* Pneumothorax;
* Use of neuromuscular blockers;
* Active tuberculosis;
* Traction devices;
* Active bleeding;
* Suspected or confirmed pulmonary embolism without prior treatment within 24 hours;
* Presence of a large mass in the right and/or left hemithorax;
* History of cardiopulmonary arrest within the past 24 hours under neuroprotection;
* In the total weaning phase from IMV and/or tracheostomy and/or enteral feeding tube and/or scheduled CT scan within the next 6 hours;
* Intolerance to the TLA test (SpO₂ drop <92% or ≥20% from baseline, need for FiO₂ increase >50% or ≥20% from baseline, need for PEEP increase, or hemodynamic instability within the first 5 minutes of lateralization testing);
* Those who refuse to provide consent, as determined by the legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory drive parameters: Surface electromyography (sEMG) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  The respiratory drive parameter will be assessed using surface electromyographic (sEMG) activity of the respiratory muscles, including the diaphragm and parasternal intercostals, expressed in microvolts (µV) (Silva Junior et al., 2023).
  Data are given in:
  • µV: Microvolts Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral Lateralization Therapy.
Respiratory drive parameter: P0.1 (airway occlusion pressure during the first 100 ms of the inspiratory effort) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes(6 hour 10 minutes)
  The respiratory drive parameter will be assessed by P0.1(airway occlusion pressure during the first 100ms of the inspiratory effort,cmH₂O).P0.1 is the drop in airway pressure within 100 ms after the onset of inspiration and is considered a reliable, fast, and feasible bedside marker.The following values are considered: Normal: 1.5-3.5 cmH₂O; Low: <1.0 cmH₂O(hypostimulated); High:>4.0 cmH₂O (hyperstimulated)(CHEN et al.,2023).
  Data are given in: cmH₂O: centimeters of water Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes Bilateral.
Respiratory drive parameters: Pmus (estimated inspiratory muscle pressure) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  The respiratory drive will be assessed using Pmus (estimated inspiratory muscle pressure). Pmus is derived from the airway pressure drop during a brief inspiratory occlusion and reflects inspiratory effort. Reference ranges: Pmus < 5 cmH₂O indicates over-assistance/low drive; Pmus ≤ 10 cmH₂O represents the diaphragmatic protection zone; Pmus > 13-15 cmH₂O indicates excessive effort (Dianti, Bertoni ;Goligher, 2020).
  Data are given in:
  •cmH₂O: centimeters of water
  Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral
Pulmonary ventilation: Ventilation Impedance Change (ΔZ) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  ΔZ will be quantified using electrical impedance tomography (EIT). ΔZ represents the sum of impedance changes of all pixels within a predefined region of interest (ROI), corresponding to regional tidal ventilation. ROIs will include right anterior, left anterior, right posterior, and left posterior lung regions, and will also be categorized as dependent or non-dependent lung areas. Data will be expressed in arbitrary units (a.u.).
  Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral Lateralization Therapy.
Pulmonary aeration: End-Expiratory Lung Impedance Change (ΔEELZ) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  ΔEELZ will be assessed using electrical impedance tomography (EIT). ΔEELZ corresponds to the aggregate end-expiratory impedance (sum of pixel values) within each ROI, representing changes in end-expiratory lung volume. ROIs will include right anterior, left anterior, right posterior, and left posterior lung regions, grouped as dependent or non-dependent areas. Data will be expressed in arbitrary units (a.u.).
  Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral Lateralization Therapy.

SECONDARY OUTCOMES:
Mechanical response associated with respiratory drive: Diaphragmatic excursion | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  Diaphragmatic excursion will be assessed by ultrasonography using a convex transducer placed along the right mid-clavicular line, using the liver as an acoustic window. The procedure follows established ICU protocols and can be performed without ventilator disconnection. In this study, ventilation will remain connected, and diaphragmatic excursion will be quantified in millimeters (mm) (Santana et al., 2020).
  Data are given in: mm: Millimeters. Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral.
Mechanical response related to respiratory effort and lung stress: Dynamic transpulmonary driving pressure | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  Dynamic transpulmonary driving pressure (cmH₂O) will assess the mechanical response to respiratory effort and lung stress. It is derived from the same expiratory occlusion maneuver used for Pmus, applying a correction formula to isolate lung distension. This provides a non-invasive measure of dynamic lung stress during ventilation. Recent studies have targeted values between 15 and 20 cmH₂O (Dianti et al., 2022).
  Data are given in: cmH₂O: centimeters of water
  Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral.
Driving Pressure (cmH₂O) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 minutes (6 hour 10 minutes)
  Driving pressure will be assessed using ventilator-derived parameters during mechanical ventilation to estimate lung stress under different body angulations and lateralization strategies. Driving pressure will be calculated as the difference between plateau pressure (Pplat) and positive end-expiratory pressure (PEEP), according to the formula: Driving Pressure = Pplat - PEEP.
  Data will be expressed in: cmH₂O (centimeters of water). Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral Lateralization Therapy.
Respiratory System Compliance (mL/cmH₂O) | Unilateral: 140 minutes (2 hours and 20 minutes) Bilateral: 370 minutes (6 hours and 10 minutes)
  Respiratory system compliance will be evaluated using ventilator-derived parameters to assess lung distensibility during different body angulations and lateralization strategies under mechanical ventilation.
  Respiratory system compliance will be calculated as the ratio between tidal volume (VT) and driving pressure, according to the formula:
  Compliance = VT/ (plateau press - PEEP).
  Data will be expressed in: cmH₂O (centimeters of water). Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral Lateralization Therapy.
Airway Resistance (cmH₂O/L/s) | Unilateral: 140 minutes (2 hours and 20 minutes) Bilateral: 370 minutes (6 hours and 10 minutes)
  Airway resistance will be measured using ventilator-derived parameters to evaluate airflow resistance during mechanical ventilation across different body angulations and lateralization strategies.
  Calculated as the difference between peak inspiratory pressure (Ppeak) and plateau pressure (Pplat) divided by inspiratory flow, according to the formula:
  Airway Resistance = (Ppeak - Pplat) / Inspiratory Flow
  Data will be expressed in: cmH₂O (centimeters of water). Measurements will be performed during the first and last 5 minutes of each body angulation. Unilateral: 140 minutes | Bilateral: 370 minutes. Following the sequence: Semi-seated 30°/20 minutes, Supine 0°/5 minutes, 15°/20 minutes, 30°/20 minutes, 15°/20 minutes, Supine 0°/5 minutes, and Semi-seated 30°/20 minutes, totaling 70 minutes per sequence plus 60 minutes of washout between sequences. This results in 140 minutes for patients undergoing Unilateral Lateralization Therapy and 370 minutes for patients undergoing Bilateral
Arterial pH | Baseline; immediately after Sequence 1; immediately after Sequence 2. Unit: pH units.
  Arterial pH measured from arterial blood gas (ABG) analysis at predefined time points: baseline (prior to the first intervention), immediately after completion of Sequence 1, and immediately after completion of Sequence 2.
  Unit: pH units.
Partial pressure of oxygen (PaO₂) | Baseline; immediately after Sequence 1; immediately after Sequence 2.
  Arterial PaO₂ measured via arterial blood gas at baseline, immediately after Sequence 1, and immediately after Sequence 2. Values obtained from arterial blood samples analyzed by standard blood gas analyzer.
  Unit: mmHg.
Partial pressure of carbon dioxide (PaCO₂) | Baseline; immediately after Sequence 1; immediately after Sequence 2.
  Arterial PaCO₂ measured via arterial blood gas at baseline, immediately after Sequence 1, and immediately after Sequence 2.
  Unit: mmHg.
Bicarbonate (HCO₃-) | Baseline; immediately after Sequence 1; immediately after Sequence 2.
  Arterial bicarbonate (HCO₃-) concentration obtained from arterial blood gas analysis at baseline, immediately after Sequence 1, and immediately after Sequence 2.
  Unit: mEq/L.
Lactate | Baseline; immediately after Sequence 1; immediately after Sequence 2.
  Arterial lactate concentration obtained from arterial blood gas or arterial blood sample at baseline, immediately after Sequence 1, and immediately after Sequence 2.
  Unit: mmol/L.
Base Excess (BE) | Baseline; immediately after Sequence 1; immediately after Sequence 2.
  Base excess determined from arterial blood gas analysis at baseline, immediately after Sequence 1, and immediately after Sequence 2.
  Unit: mEq/L.
PaO₂/FiO₂ ratio | Baseline; immediately after Sequence 1; immediately after Sequence 2.
  PaO₂/FiO₂ ratio calculated from arterial PaO₂ and the fraction of inspired oxygen (FiO₂) at baseline, immediately after Sequence 1, and immediately after Sequence 2. FiO₂ will be recorded at the time of each arterial blood gas sampling.
  Ratio (unitless).
Pulmonary Severity - LUS Score (Lung Ultrasound Score) | Baseline, immediately after Sequence 1, and immediately after Sequence 2.
  Pulmonary severity will be assessed using lung ultrasound (LUS), quantified by the Lung Ultrasound Score (LUS Score). Assessments will occur at three predefined time points: baseline (prior to the first intervention), immediately after the completion of Sequence 1, and immediately after the completion of Sequence 2.
  Pulmonary aeration will be classified according to standardized LUS Score criteria Mongodi, Silvia et al. Anesthesiology, 2021.
  Score 0: Normal lung pattern; up to two isolated B-lines. Score 1: Up to four B-lines, indicating mild loss of aeration. Score 2: More than four B-lines or confluent B-lines, indicating moderate loss of aeration.
  Score 3: Consolidations with coarse artifacts and pleural irregularities, indicating severe loss of aeration.
  Outcome Units: Ordinal scale (0 to 3 per region) and total summed score.
Hemodynamic Instability Events | At any time during the intervention and immediately after completion.
  Number of hemodynamic instability episodes defined by sustained Mean Arterial Pressure (MAP) < 60 mmHg or > 120 mmHg, each lasting more than 10 minutes, recorded throughout the intervention period. Unit: Number of events
Psychomotor Agitation - Richmond Agitation-Sedation Scale (RASS Score) | Unilateral: 140 minutes (2 hour 20 minutes) | Bilateral: 370 min (6 hour 10 minutes)
  Psychomotor agitation or sedation will be assessed using the Richmond Agitation-Sedation Scale (RASS) during each predefined body position and angulation throughout the therapy sequence.
  The RASS score ranges from -5 (unarousable) to +4 (combative), with higher positive scores indicating greater agitation and more negative scores indicating deeper levels of sedation.
  During each body position and angulation within the intervention sequence, assessed at the end of each positioning period, including:
  Semi-seated 30° (20 minutes) Supine 0° (5 minutes) Lateralization 15° (20 minutes) Lateralization 30° (20 minutes) Lateralization 15° (20 minutes) Supine 0° (5 minutes) Semi-seated 30° (20 minutes), for a total of 70 minutes per sequence, with a 60-minute washout period between sequences.
Oxygenation and Hypoxemia Events (SpO₂ Monitoring + Hypoxemia Criteria) | Continuous monitoring; events recorded at any time during the intervention.
  Continuous monitoring of peripheral oxygen saturation (SpO₂) during each therapy session.
  Any episode meeting one or more of the following hypoxemia criteria will be recorded:
  * SpO₂ < 92%, or > 20% decrease from baseline;
  * Need to increase FiO₂ > 50% or > 20% above baseline;
  * Need to increase PEEP;
  * Associated hemodynamic instability (including changes in PAM according to predefined limits).
  All events will be documented throughout the intervention. Unit: Number of events.
Unplanned Removal of Devices | During the intervention.
  Occurrence of unplanned removal of tubes or catheters during therapy (e.g., endotracheal tube, feeding tube, urinary catheter). Unit: Number of events.
Serious Adverse Events | During the intervention.
  Occurrence of pneumothorax, cardiopulmonary arrest, or any event requiring emergency interruption or modification of therapy. Unit: Number of events.

OTHER OUTCOMES:
Clinical Severity - SAPS 3 (Baseline) | Baseline (pre-intervention).
  Baseline clinical severity will be assessed using the Simplified Acute Physiology Score 3 (SAPS 3). This score provides a standardized measure of acute illness severity based on physiological, laboratory, and clinical variables collected within the first hours of ICU admission. SAPS 3 generates a total score typically ranging from 0 to 217, with higher scores indicating greater severity and higher predicted mortality risk (Salluh; Soares, 2014). The score will be recorded once before any intervention and used solely for sample characterization and stratification.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Fernandes Ferreira da Silva Júnior, MSc, Principal Investigator — Federal University of Pernambuco (UFPE) - Health-Applied Biology Graduate Program, Federal University of Pernambuco, Recife, Brazil; Shirley Lima Campos Lima Campos, PhD, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Hospital Geral Otávio de Freitas - Secretaria de Saúde de Pernambuco, Recife, Pernamu, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Participant characteristics Medical history Clinical measurements Functional results Images (USG) Adverse events
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Through study completion
Access Criteria: Individual participant data (IPD) access will be granted by the PI after request review for approval via email. It will be shared with researchers and general public of interest on the subject for descriptive analyses related to our sample. A committee of researchers will be in charge of discussing the request before approving the access.

REFERENCES:
- [Background] Salluh JI, Soares M. ICU severity of illness scores: APACHE, SAPS and MPM. Curr Opin Crit Care. 2014 Oct;20(5):557-65. doi: 10.1097/MCC.0000000000000135. PMID 25137401
- [Background] Dianti J, Bertoni M, Goligher EC. Monitoring patient-ventilator interaction by an end-expiratory occlusion maneuver. Intensive Care Med. 2020 Dec;46(12):2338-2341. doi: 10.1007/s00134-020-06167-3. Epub 2020 Jul 4. No abstract available. PMID 32623476
- [Background] Chen H, Liang M, He Y, Teboul JL, Sun Q, Xie J, Yang Y, Qiu H, Liu L. Inspiratory effort impacts the accuracy of pulse pressure variations for fluid responsiveness prediction in mechanically ventilated patients with spontaneous breathing activity: a prospective cohort study. Ann Intensive Care. 2023 Aug 17;13(1):72. doi: 10.1186/s13613-023-01167-0. PMID 37592166
- [Background] Silva Junior EFFD, Campos SL, Leite WS, Melo PVS, Lins RAC, Araujo MDGR, Guerino MR. Surface electromyography signal processing and evaluation on respiratory muscles of critically ill patients: A systematic review. PLoS One. 2023 Apr 27;18(4):e0284911. doi: 10.1371/journal.pone.0284911. eCollection 2023. PMID 37104255
- [Background] Costa LSP, Reinaux CMA, Junior EFFS, Leite WS, Brandao DC, de Andrade AD, Roldan R, Morais CCA, Campos SL. Physiology of body lateralization on regional lung ventilation and lung volumes in healthy subjects: Within-subjects design. PLoS One. 2025 Oct 30;20(10):e0335622. doi: 10.1371/journal.pone.0335622. eCollection 2025. PMID 41166369
- [Background] Zack MB. Pectoriloquy, a retrospective analysis. Chest. 2009 Jan;135(1):8-9. doi: 10.1378/chest.08-2261. No abstract available. PMID 19136401
- [Background] Vedrenne-Cloquet M, Ito Y, Hotz J, Klein MJ, Herrera M, Chang D, Bhalla AK, Newth CJL, Khemani RG. Phenotypes based on respiratory drive and effort to identify the risk factors when P0.1 fails to estimate ∆PES in ventilated children. Crit Care. 2024 Oct 4;28(1):325. doi: 10.1186/s13054-024-05103-x. PMID 39367452
- [Background] Umbrello M, Formenti P, Longhi D, Galimberti A, Piva I, Pezzi A, Mistraletti G, Marini JJ, Iapichino G. Diaphragm ultrasound as indicator of respiratory effort in critically ill patients undergoing assisted mechanical ventilation: a pilot clinical study. Crit Care. 2015 Apr 13;19(1):161. doi: 10.1186/s13054-015-0894-9. PMID 25886857
- [Background] Suttapanit K, Wongkrasunt S, Savatmongkorngul S, Supatanakij P. Ultrasonographic evaluation of the diaphragm in critically ill patients to predict invasive mechanical ventilation. J Intensive Care. 2023 Sep 19;11(1):40. doi: 10.1186/s40560-023-00690-3. PMID 37726832
- [Background] Schifino G, Vega ML, Pisani L, Prediletto I, Catalanotti V, Comellini V, Bassi I, Zompatori M, Ranieri MV, Nava S. Effects of non-invasive respiratory supports on inspiratory effort in moderate-severe COVID-19 patients. A randomized physiological study. Eur J Intern Med. 2022 Jun;100:110-118. doi: 10.1016/j.ejim.2022.04.012. Epub 2022 Apr 22. PMID 35483993
- [Background] ROSA, Jéssica dos Santos Pereira et al. Impacts in the Respiratory Mechanics of the Ventilator Hyperinsuflation in the Flow Bias Concept: a Narrative Review. Journal of Health Sciences, v. 21, n. 3, p. 250-254, 2019.
- [Background] Roesthuis LH, van der Hoeven JG, van Hees HWH, Schellekens WM, Doorduin J, Heunks LMA. Recruitment pattern of the diaphragm and extradiaphragmatic inspiratory muscles in response to different levels of pressure support. Ann Intensive Care. 2020 May 29;10(1):67. doi: 10.1186/s13613-020-00684-6. PMID 32472272
- [Background] Dos Santos Rocha A, Diaper J, Balogh AL, Marti C, Grosgurin O, Habre W, Petak F, Sudy R. Effect of body position on the redistribution of regional lung aeration during invasive and non-invasive ventilation of COVID-19 patients. Sci Rep. 2022 Jun 30;12(1):11085. doi: 10.1038/s41598-022-15122-9. PMID 35773299
- [Background] Pearce AK, McGuire WC, Elliott AR, Goligher EC, Prisk GK, Butler JP, Malhotra A. Impact of Supine Versus Semirecumbent Body Posture on the Distribution of Ventilation in Acute Respiratory Distress Syndrome. Crit Care Explor. 2023 Dec 1;5(12):e1014. doi: 10.1097/CCE.0000000000001014. eCollection 2023 Dec. PMID 38053751
- [Background] Kubota S, Hashimoto H, Yoshikawa Y, Hiwatashi K, Ono T, Mochizuki M, Naraba H, Nakano H, Takahashi Y, Sonoo T, Nakamura K. Effects of mechanical insufflation-exsufflation on ventilator-free days in intensive care unit subjects with sputum retention; a randomized clinical trial. PLoS One. 2024 May 2;19(5):e0302239. doi: 10.1371/journal.pone.0302239. eCollection 2024. PMID 38696429
- [Background] Huerta MDR, Giralt JAS, Diez-Fernandez A, Alonso MJR, Montes N, Suarez-Sipmann F. Effects of routine postural repositioning on the distribution of lung ventilation and perfusion in mechanically ventilated patients. Intensive Crit Care Nurs. 2025 Apr;87:103952. doi: 10.1016/j.iccn.2025.103952. Epub 2025 Jan 25. PMID 39864264
- [Background] Gong S, Lian H, Ding X, Wang X; Chinese Critical Ultrasound Study Group (CCUSG). High Respiratory and Cardiac Drive Exacerbate Secondary Lung Injury in Patients With Critical Illness. J Intensive Care Med. 2025 Mar;40(3):231-238. doi: 10.1177/08850666231222220. Epub 2024 Jan 3. PMID 38173252
- [Background] Franchineau G, Jonkman AH, Piquilloud L, Yoshida T, Costa E, Roze H, Camporota L, Piraino T, Spinelli E, Combes A, Alcala GC, Amato M, Mauri T, Frerichs I, Brochard LJ, Schmidt M. Electrical Impedance Tomography to Monitor Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2024 Mar 15;209(6):670-682. doi: 10.1164/rccm.202306-1118CI. PMID 38127779
- [Background] Cherniack NS, Lederer DH, Altose MD, Kelsen SG. Occlusion pressure as a technique in evaluating respiratory control. Chest. 1976 Jul;70(1 Suppl):137-41. doi: 10.1378/chest.70.1_supplement.137. No abstract available. PMID 939129
- [Background] Caetano DS, Morais CC, Leite WS, Lins RAC, Medeiros KJ, Cornejo RA, de Andrade AD, Campos SL, Brandao DC. Electrical Impedance Tomographic Mapping of Hypoventilated Lung Areas in Intubated Patients With COVID-19. Respir Care. 2023 Jun;68(6):773-776. doi: 10.4187/respcare.10261. Epub 2023 Apr 25. No abstract available. PMID 37185111
- [Background] Brito ALA, Ferreira ACA, Costa LSP, Silva Junior EFF, Campos SL. Effect of Continuous Lateral Rotation Therapy on Clinical Outcomes in Mechanically Ventilated Critically Ill Adults. Respir Care. 2024 Nov 18;69(12):1592-1606. doi: 10.4187/respcare.11781. PMID 38744476
- [Background] Bonczynski GS, Novo JS, Dias AS, Martins LFG, Naue WDS, Volpe MS, Junior LAF. Ventilator hyperinflation associated with flow bias optimization in the bronchial hygiene of mechanically ventilated patients. Heart Lung. 2024 Mar-Apr;64:31-35. doi: 10.1016/j.hrtlng.2023.10.011. Epub 2023 Nov 21. PMID 37988854
- [Background] Bertoni M, Telias I, Urner M, Long M, Del Sorbo L, Fan E, Sinderby C, Beck J, Liu L, Qiu H, Wong J, Slutsky AS, Ferguson ND, Brochard LJ, Goligher EC. A novel non-invasive method to detect excessively high respiratory effort and dynamic transpulmonary driving pressure during mechanical ventilation. Crit Care. 2019 Nov 6;23(1):346. doi: 10.1186/s13054-019-2617-0. PMID 31694692
- [Background] American Association for Respiratory Care. AARC Clinical Practice Guidelines. Endotracheal suctioning of mechanically ventilated patients with artificial airways 2010. Respir Care. 2010 Jun;55(6):758-64. PMID 20507660
- [Background] Alcala GC, Ekkapat G, Medeiros KJ, Morais CCA, Xin Y, Giammatteo V, Bruno G, Nova A, Wanderley H, Buhl T, Victor M, Gaulton TG, La Vita CJ, Amato MBP, Ceradda M, Berra L, Ribeiro De Santis Santiago R. Monitoring Lung Function with Electrical Impedance Tomography in the Intensive Care Unit. J Vis Exp. 2024 Sep 6;(211). doi: 10.3791/66756. PMID 39311582
- Available data/document: Study Protocol: Multicare: Bed for protocol — https://drive.google.com/file/d/1tTjIHQ18FQa7SDYQpLIKStPNh8LqN09o/view?usp=sharing — The Multicare: Bed for Protocol is used to standardize therapeutic positioning, ensuring precision and safety in evaluating the postural effects on lung aeration and respiratory drive